CLINICAL TRIAL: NCT00126958
Title: Cost-Effectiveness of Follow-up of Patients With Superficial Bladder Cancer
Brief Title: Cost-Effectiveness in Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Reinier de Graaf Groep (Other); Sint Franciscus Gasthuis (Other); Vlietland Ziekenhuis (Other); Medisch Centrum Rijnmond-Zuid, Netherlands (Other Government); Havenziekenhuis (Other); Albert Schweitzer Hospital, Netherlands (Unknown); Ikazia Hospital, Rotterdam (Other); Leiden University Medical Center (Other)
Other Study IDs: *ZON-MW 945-02-046*
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2005-08

CONDITIONS: Bladder Cancer
Keywords: superficial urothelial cell carcinoma; urinary analysis; Loss of heterozygosity; FGFR3 mutation; follow-up
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Urinary Sediment Analysis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: urinary analysis

SUMMARY:
This randomized clinical multicentre trial aims to evaluate the efficacy of microsatellite analysis on voided urine to detect tumour recurrences in the follow-up of patients with superficial urothelialcell carcinoma (UCC). Further, this study aims to identify subgroups of patients with a low risk of tumour recurrence using clinico-pathologic tumour characteristics in combination with a genetic marker (FGFR3 gene), such that the frequency of follow-up contact can be reduced. The overall objective is to reduce the frequency of cystoscopy during follow-up in patients with superficial UCC, leading to an improvement in quality of life at equal or lower costs. This study evaluates the cost-effectiveness of follow-up in bladder cancer.

DETAILED DESCRIPTION:
The randomized clinical study consists of two intervention arms. The control arm consists of a conventional follow-up based on regular monitoring for urinary bladder UCC recurrences by cystoscopy. In the test arm a proportion of the cystoscopies is replaced by microsatellite analysis on voided urine. Both arms will be stratified for clinical and pathological tumour parameters as well as for the mutation status of the prognostic FGFR3 gene mutation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with resectable pT1 or pTa, grade G1-G2 transitional cell carcinoma of the bladder which is biopsy proven

Exclusion Criteria:

* Patients who present or presented with a transitional cell carcinoma of the bladder, stage pT2 or more invasive, or carcinoma in situ (CIS) and/or G3 diagnosed in history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2002-07; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Th. van der Kwast, Prof PhD MD, Principal Investigator — Erasmus MC, JNI; E.C. Zwarthoff, Ph.D, Principal Investigator — Erasmus MC, JNI